CLINICAL TRIAL: NCT04263493
Title: Delayed Loading Following Repair of a Ruptured Achilles Tendon - a Randomized Controlled Trial
Brief Title: Delayed Loading Following Repair of a Ruptured Achilles Tendon
Acronym: DELOAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Rikke Høffner, PhD student, MSc, PT, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01012020
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles Tendon Surgery
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early mobilization (loading) (Active Comparator): This constitutes the currently accepted regime and is therefore considered the control group.
  Cast/orthopedic boot for 6 weeks No weight bearing: week 0-2 Partiel weightbearing from week 3 Full weightbearing from week 7 ROM exercises 5 times a day from week 3
  Interventions: Other: Rehabilitation (physiotheraphy)
- Delayed mobilization (loading) (Experimental): Loading of the Achilles tendon is delayed for 6 weeks. Cast/orthopedic boot for 12 weeks No weight bearing: week 0-6 Partiel weightbearing from week 7 Full weightbearing from week 13 ROM exercises 5 times a day from week 3
  Interventions: Other: Rehabilitation (physiotheraphy)

INTERVENTIONS:
Other: Rehabilitation (physiotheraphy) — Time of loading, range of motion exercises, strength training

SUMMARY:
The purpose of the study is to investigate if delayed loading following surgical treated Achilles tendon rupture influence the clinical outcome and muscle and tendon structure after one year.

The investigators hypothesize that delaying the gradual introduction of loading in the initial 26 weeks may reduce the heel-rise deficit (primary outcome) and thus improve the clinical outcome one year after surgery (primary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a traumatic, complete mid-substance Achilles tendon
* No contraindications for MRI
* Presented within 14 days from injury
* Adult (18 to 60 years)
* Understand Danish
* Manage transport to/from the hospital on their own

Exclusion Criteria:

* Other injuries affecting their lower limb functions
* Prior Achilles tendon Rupture
* Smoking
* Systemic diseases influencing tendon healing
* Anticoagulation treatment
* Inability to follow rehabilitation or complete follow-ups
* Immunosuppressive treatment including systematic corticosteroid treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Heel-rise test | One-year follow-up
  Heel-rise height deficit on the injured side relative to the uninjured side

SECONDARY OUTCOMES:
Tendon length and cross-sectional area | 1 week, 3 months, 6 months and 1 year
  MRI will be used to measure free tendon length, tendon cross-sectional area and tendon length up to the gastrocnemius insertion.
The Achilles tendon rupture score (ATRS) | Recall before injury and 1 year
  The Achilles tendon rupture score questionnaire is a patient-reported outcome with a possible score from 1-100, where higher scores mean a better outcome.
Muscle fascicle length and doppler activity in the tendon | 2 weeks, 3 months, 6 months and 1 year
  Muscle fascicle length and doppler activity in the tendon will be measured with ultrasonography
Isokinetic plantar flexion muscle strength | 1 year
  The Biodex is used to obtain isokinetic plantar flexion muscle strength during maximal contractions.
Physical activity level | Recall before injury and 1 year
  A questionnaire is used to measure the physical activity level (including type of activity) of the participants.
Heel-rise work | 6 months and 1 year
  An instrumented heel-rise test will be conducted to measure work capacity
The Achilles tendon resting angle (ATRA) | 2 weeks, 3 months, 6 months and 1 year
  Achilles tendon resting angle will be measured using a standard goniometer. Measurements will be obtained with the knee flexed and extended.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Magnusson, Professor, Principal Investigator — Institute of Sportsmedicine
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoeffner R, Svensson RB, Gillani SZ, Linden FH, Magnusson SP. Morphological Changes One Year After Achilles Tendon Rupture Repair: A Comparison of Loading Strategies. Transl Sports Med. 2025 Sep 28;2025:1778630. doi: 10.1155/tsm2/1778630. eCollection 2025. PMID 41059465
- [Derived] Hoeffner R, Agergaard AS, Svensson RB, Cullum C, Mikkelsen RK, Konradsen L, Krogsgaard M, Boesen M, Kjaer M, Magnusson SP. Tendon Elongation and Function After Delayed or Standard Loading of Surgically Repaired Achilles Tendon Ruptures: A Randomized Controlled Trial. Am J Sports Med. 2024 Mar;52(4):1022-1031. doi: 10.1177/03635465241227178. Epub 2024 Feb 14. PMID 38353060

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT04263493/Prot_SAP_000.pdf